CLINICAL TRIAL: NCT05824936
Title: Enhanced Community-Based Asthma Monitoring Through Novel Technology
Acronym: EMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Abigail Strang, PI/MD, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2002602; P20GM144270 (NIH)
Record Dates: First submitted 2023-03-20; First posted 2023-04-24 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Asthma in Children
Keywords: asthma; spirometry; telehealth
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: 15 participants will be enrolled in single-group pilot study to measure acceptability, feasibility, and accessibility of mobile spirometry for asthma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot study arm for technology-enhanced asthma intervention (Experimental): All participants will be in the pilot arm for technology-enhanced intervention program.
  Interventions: Behavioral: Pilot study arm for technology-enhanced asthma intervention

INTERVENTIONS:
Behavioral: Pilot study arm for technology-enhanced asthma intervention — Participants will be enrolled in a remote monitoring program using monthly remote study visits which will include the use of a mobile spirometer (device for testing lung function). Participants will complete monthly remote study visits visits using telehealth platform and will complete lung function testing during the visit using a mobile spirometer as well as remote study measures.

SUMMARY:
The goal of this pilot interventional study is to learn about the implementation of a home monitoring program (using remote study visits and lung function testing) in children with asthma.

The main questions to answer are:

1. Do participants find the program to be feasible, acceptable and accessible?
2. What factors are associated with completion of the program?
3. Does the program have an effect on asthma control and daytime sleepiness?

DETAILED DESCRIPTION:
The primary objective of the proposed study is to pilot test implementation of a protocol for enhanced asthma monitoring using novel technology, including mobile spirometry and remote study visits, for rural and medically underserved children with persistent asthma in Delaware and to determine its feasibility, acceptability, and accessibility.

Additionally, the proposed study aims to explore patient and family demographic characteristics and social factors associated with successful completion of the program and to explore the preliminary effect of the enhanced asthma monitoring program on asthma control and sleepiness as a measure of daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* Followed by a Primary Care Practice meeting HRSA rural or medically underserved designation status
* Diagnosis of persistent asthma: on at least 1 controller/ preventative medication for asthma
* Ability to follow directions and perform study measures, including in-office spirometry at initial visit
* Access to mobile device with internet connectivity to connect to telehealth visit and mobile spirometer application

Exclusion Criteria:

* Significant cardiopulmonary disease other than asthma (Examples: Cystic Fibrosis, complex congenital heart disease)
* Non-English Speaking

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 15 participants enrolled in pilot intervention
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Retention %)
Description: Feasibility will be evaluated by calculating retention rates at week 24.
Time Frame: 24 weeks
Population: Participants who completed the pilot through final study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 15
Participants | 14

2. Primary Outcome: Acceptability
Description: To measure acceptability, the study-specific Satisfaction and Usability Survey will be used and assessed at item-level. The percentage (%) of participants who respond "agree" or "strongly agree" to each item will be measured.
Time Frame: 24 weeks
Population: Results of Satisfaction and Usability Survey for 12 participants who completed the pilot and also completed this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 12
Participants
  It was easy to use | 12
  It was convenient to use | 12
  The time spent was just about right. | 12
  The introduction and training was enough. | 12
  I would recommend the program to others. | 12
  It helped me change my asthma habits. | 11
  It helped me to understand the importance of following my asthma plan. | 10
  It helped me to understand how to control my asthma. | 10
  It helped me to manage my asthma in a way that I could not have done myself. | 10
  It helped me to understand my asthma better. | 11

3. Primary Outcome: Accessibility
Description: The frequency (%) of any technical or connectivity issues at each visit will be recorded throughout the study.
Time Frame: 24 weeks
Population: Remote visits (5 total) of 14 participants who completed pilot were analyzed for technical concerns.
Measure: Count of Units; unit: Remote study visits
Units Other Than Participants: Remote study visits
Groups:
- Pilot Study Arm for Technology-enhanced Asthma Intervention: All participants who completed the pilot arm.
  Pilot study arm for technology-enhanced asthma intervention: Participants will be enrolled in a remote monitoring program using monthly remote study visits which will include the use of a mobile spirometer (device for testing lung function). Participants will complete monthly remote study visits visits using telehealth platform and will complete lung function testing during the visit using a mobile spirometer as well as remote study measures.
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 14
Number analyzed (Remote study visits) | 70
Remote study visits
  Visits with Technical Challenges | 9
  Visits without technical challenges | 61

4. Secondary Outcome: Explore the Preliminary Effectiveness of the Pilot Program on Asthma Control.
Description: The asthma control test (ACT) will be completed at each study visit. This measure rates asthma symptoms from 5-25 with 5 being the lowest (poorest) asthma control and 25 being the highest (optimal) asthma control.
Time Frame: Baseline and Week 24
Population: ACT of 14 participants who completed the pilot were analyzed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 14
score on a scale
  Baseline ACT -Week 0 (median) | 23 [14 to 25]
  Final ACT- Week 24 (median) | 22 [12 to 25]

5. Secondary Outcome: Explore the Preliminary Effectiveness of the Pilot Program on Daytime Sleepiness.
Description: The Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) will be completed at each study visit. This measure rates sleepiness with scores of 0-24 with 0 being the lowest degree of daytime sleepiness and 24 being the highest (sleepiest).
Time Frame: Baseline and Week 24
Population: ESS-CHAD scores of all participants who completed the pilot.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
Number analyzed (Participants) | 14
score on a scale
  Baseline Week 0 ESS-CHAD (Median) | 6 [0 to 14]
  Final- Week 24 ESS-CHAD (median) | 4 [0 to 15]

6. Secondary Outcome: Explore Patient and Family-related Demographic Characteristics and Psychosocial Factors Associated With Successful Completion of the Intervention.
Description: The study-specific demographic and psychosocial assessment tool will be completed at the baseline visit. Descriptive and comparative statistics will be employed to characterize participant-specific demographic factors which may be associated with study completion at item-level.
Time Frame: 24 weeks
Population: Characteristics of participants who completed pilot were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Completed Pilot Study Arm: Participants in study arm who successfully completed the pilot.
- Participants Who Did Not Complete Pilot: Participants who did not complete pilot.
Arm/Group | Completed Pilot Study Arm | Participants Who Did Not Complete Pilot
Number analyzed (Participants) | 14 | 1
Participants
  Ethnicity: Hispanic | 3 | 0
  Ethnicity: Non-Hispanic | 11 | 1
  Sex: Male | 4 | 1
  Sex: Female | 10 | 0
  Race: White | 7 | 0
  Race: Black or African-American | 4 | 1
  Race: More than one race | 3 | 0

7. Secondary Outcome: Explore Asthma-related Factors Associated With Successful Completion of the Intervention (Oral Steroid Usage)
Description: Asthma-related factors associated with successful completion of the intervention will be analyzed and compared to participants who do not complete the intervention. Courses of oral steroids in the prior 6 months were calculated based on participant survey results.
Time Frame: Baseline
Population: Asthma-related baseline characteristics of participants who completed vs. did not complete the pilot were compared and analyzed.
Measure: Median (Full Range); unit: Courses
Groups:
- Participants Who Did Not Complete the Pilot: Participants who did not complete the pilot (drop out).
Arm/Group | Completed Pilot Study Arm | Participants Who Did Not Complete the Pilot
Number analyzed (Participants) | 14 | 1
Courses | 1 [0 to 10] | 0 [0 to 0]

8. Secondary Outcome: Explore Asthma-related Factors Associated With Successful Completion of the Intervention (ER Visits)
Description: Asthma-related factors associated with successful completion of the intervention will be analyzed and compared to participants who do not complete the intervention. Number of ER visits were calculated based on survey results
Time Frame: Baseline
Population: as for outcome 7
Measure: Median (Full Range); unit: ER visits
Arm/Group | Completed Pilot Study Arm | Participants Who Did Not Complete the Pilot
Number analyzed (Participants) | 14 | 1
ER visits | 1 [0 to 10] | 0 [0 to 0]

9. Secondary Outcome: Explore Asthma-related Factors Associated With Successful Completion of the Intervention (Hospital Admissions)
Description: Asthma-related factors associated with successful completion of the intervention will be analyzed and compared to participants who do not complete the intervention. Hospital admissions were calculated based on survey results.
Time Frame: Baseline
Population: as for outcome 7
Measure: Median (Full Range); unit: Admissions
Arm/Group | Completed Pilot Study Arm | Participants Who Did Not Complete the Pilot
Number analyzed (Participants) | 14 | 1
Admissions | 0 [0 to 5] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pilot Study Arm for Technology-enhanced Asthma Intervention
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT05824936/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT05824936/ICF_001.pdf